CLINICAL TRIAL: NCT02857907
Title: Anti-thymocyte Globulin-induced Immune Senescence
Acronym: SIGAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2010/15
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Kidney transplantation; Immunosuppressive treatment
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ATG group: Patients who received T cell depleting ATG therapy (blood sample one year after transplantation)
  Interventions: Other: Blood sample
- anti-CD25 group: Patients who received nondepleting anti-CD25 (blood sample one year after transplantation)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample is performed one year after kidney transplantation.

SUMMARY:
The aim of the study is to investigate the impact of Anti-Thymocyte Globulin (ATG) on immune senescence. Markers of immune senescence expression is assessed in a prospective cohort of renal transplant recipients the day of transplantation and one year after renal transplantation.

DETAILED DESCRIPTION:
The anti-thymocyte globulin (ATG) are used in the prevention and treatment of acute rejection in organ transplantation. They are at the origin of a brutal CD4 lymphocyte depletion followed by a gradual recovery of the lymphocyte pool. Nevertheless, CD4 lymphopenia can persist in some patients.

SIGAL study aims to characterize the immune responses of lymphopenic patients (after administration of ATG) in order to identify possible similarities with immunosenescence.The immunosenescence is a complex and profound remodeling of the immune system during life. It is mainly due to thymic involution and repeated antigenic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to understand the reason of the study
* Signature of informed consent
* Patient who are waiting renal transplant

Exclusion Criteria:

* Inability to understand the reasons for the study; psychiatric disorders
* Any history in the last 2 years of immunosuppressive therapy (except steroids)
* History of cancer (except skin cancer) or treated hematological malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients awaiting kidney transplantation, followed at Besançon University Hospital and who have given their consent for the conservation of cells for a study of the immune system in kidney transplant patients.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Percentage of senescent lymphocytes | One year after kidney transplantation
  Flow cytometry analysis (7 colors) of lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Bamoulid, Doctor, Principal Investigator — CHU Besançon
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No